CLINICAL TRIAL: NCT05105269
Title: Do Working Alliance, Patient Outcome Expectations and Self-efficacy Predict Change in Pain and Disability From Treatment With a Physiotherapist for Achilles Tendinopathy
Brief Title: Managing Achilles Pain II
Acronym: MAP II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Essex (Other)
Collaborators: Chartered Society of Physiotherapy (Unknown)
Responsible Party: Sponsor
Other Study IDs: ETH2021-1779
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment from a physiotherapist — Any treatment provided by a physiotherapist e.g. exercise, advice and massage

SUMMARY:
Although some people are more at risk than others, developing a painful Achilles tendon (known as Achilles tendinopathy) can affect anyone. It is a common and disabling condition affecting walking, running and work. To reduce the pain and disability, exercise is a commonly used treatment by physiotherapists. However, success varies. This is why the proposed research is needed, to identify the factors that predict changes in pain and disability from treatment with a physiotherapist. The investigators' previous research suggests the working relationship or 'alliance' between the physiotherapist and patient, the patient's expectations, and the patient's confidence to carry out exercise might be important, but further research is needed to determine this.

The investigators have designed a multi-centre, longitudinal cohort study to assess whether working alliance, patient expectations of treatment success, and confidence to perform exercise (self-efficacy) predict changes in pain and disability from a treatment programme prescribed by a physiotherapist for Achilles tendinopathy at twelve weeks. Patients, diagnosed with Achilles tendinopathy by their treating physiotherapist, will be introduced to the study through a verbal discussion and provided with details of the study's website (www.managing-achilles-pain.com). The website provides password protected information (the participant information sheet, consent form and a questionnaire measuring clinical outcomes and the predictive factors). The participant is asked to complete the questionnaire on three occasions; baseline, six weeks later and twelve weeks after baseline.

DETAILED DESCRIPTION:
Pain related to a tendon, termed tendinopathy, can be traumatic or insidious in onset and short-lasting or persistent in nature. Tendinopathy is common musculoskeletal condition; the incidence of tendinopathy is higher than osteoarthritis, for example. Achilles tendinopathy (AT) affects both active and sedentary individuals and can be characterised by reduced activity tolerance to specific tasks that load the tendon. This results in decreased activity participation such as walking, running and working.

Current clinical guidelines recommend exercise as the first line treatment for people with Achilles tendinopathy. However, the rate and extent of improvement in pain and disability varies. This variation suggests the investigators need to understand what factors predict change so the investigators can enhance care provided. Previously it was suggested that exercise worked by improving the strength or structure of the tendon, but it has been reported that pain and disability can change without corresponding changes in strength or structure. This suggests that other factors might be important predictors.

Recent literature suggests cognitive and contextual influences such as self-efficacy, working alliance and expectations may be important factors for predicting change in pain and disability in tendinopathy and need investigation. Based on this need, high-quality research is warranted. To inform the development of this research, two recent studies have been undertaken. Firstly, a feasibility study was completed. This study aimed to understand if it was feasible to collect data using a secure website to explore the association and predictive relationship of working alliance, outcome expectations and self-efficacy with pain and disability in the management of AT. The second study was a process evaluation to gain insight into the procedures undertaken in the feasibility study. Seven patients were interviewed to discover what worked (and did not) from their perspective during the study. Based on the results from the feasibility study and the information from the interviews with patients, using this website is feasible, but the investigators have made some changes before proposing this larger study. These changes include better promotion of the study, how verbal recruitment strategies could be improved, and how communication between clinicians and researchers could be made better. Based upon this knowledge this proposal aims to understand if working alliance, patient outcome expectations and self-efficacy predict response to treatment for AT.

ELIGIBILITY:
Inclusion Criteria:

* be a minimum of 18 years old
* have access to the internet
* have an available email address
* to have support in place to understand written English if it is required
* be diagnosed with AT by their treating physiotherapist
* be undertaking treatment prescribed by a physiotherapist.

Exclusion Criteria:

* not provided informed consent
* been diagnosed with Achilles tendon tear/rupture
* received surgery to the affected Achilles tendon
* pain in the Achilles region with movements of the spine or neural tissue

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosis of Achilles tendinopathy will be based on criteria from expert consensus: local mid-portion Achilles tendon pain reproduced with load-based activity and tenderness on palpation
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale | 3 months
  The LEFS is a self-report questionnaire designed to measure physical function of people with lower extremity dysfunctions, such as AT. Twenty items covering a range of lower extremity functional activities are scored on a numerical rating scale from zero (extreme difficulty or unable to perform activity) to four (no difficulty). This provides maximum scale points of eighty, with zero representing maximum dysfunction.

SECONDARY OUTCOMES:
Numerical Pain Scale | 3 months
  The NPRS is an 11-point scale designed to measure self-reported pain intensity on a scale ranging between 0 (no pain at all) and 10 (the worst pain ever possible)

CONTACTS AND LOCATIONS:
Locations (1):
- Connect Health, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT05105269/Prot_000.pdf